CLINICAL TRIAL: NCT04415307
Title: The Efficacy and Safety of Traditional Chinese Medicine (TCM) to the Patient With Dizziness in Emergency Department
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: principal investigator leave the organization
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191250
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Dizziness
MeSH Terms: conditions — Dizziness | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Acupuncture (Experimental): Acupuncture over acupoints.
  Interventions: Other: Acupuncture
- Far-Infrared (Experimental): Far-Infrared heat-patch attachment over acupoints.
  Interventions: Other: Far-Infrared heat-patch attachment
- Combination of Acupuncture and Far-Infrared (Experimental): Acupuncture and Far-Infrared heat-patch attachment over acupoints.
  Interventions: Other: Acupuncture and Fir-Infrared heat-patch attachment
- Placebo (no Acupuncture nor Far-Infrared) (Placebo Comparator): Far-Infrared heat-patch attachment over acupoints without electric current passing.
  Interventions: Other: Far-Infrared heat-patch attachment over acupoints without electric current passing.

INTERVENTIONS:
Other: Acupuncture — Acupuncture over acupoints.
  Arms: Acupuncture
Other: Far-Infrared heat-patch attachment — Far-Infrared heat-patch attachment over acupoints.
  Arms: Far-Infrared
Other: Acupuncture and Fir-Infrared heat-patch attachment — Acupuncture and Far-Infrared heat-patch attachment over acupoints.
  Arms: Combination of Acupuncture and Far-Infrared
Other: Far-Infrared heat-patch attachment over acupoints without electric current passing. — Far-Infrared heat-patch attachment over acupoints without electric current passing.
  Arms: Placebo (no Acupuncture nor Far-Infrared)

SUMMARY:
The study is aimed in patients with persistent dizziness as the chief complaint that is treated with acupuncture or/and far-infrared heat-patch attachment intervention over the acupoints for the purpose of dizziness symptoms treatment. The research hypothesis is that the treatment over acupoints in traditional Chinese medicine is effective in treating symptoms of dizziness.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age between 20 to 80-year-old who can cooperate to the whole treatment, testing and questionnaire.
2. The chief complaint is dizziness which diagnosed by the doctor in charge of the emergency department, in together to exclude the patients with severe unstable vital signs, and then consult for help with Chinese medicine.
3. Sign the clinical trial agreement sheet.

Exclusion Criteria:

1. Inacceptable to the research content
2. Unable to complete the study process
3. Unwilling to cooperate with acupuncture and other treatments
4. Abnormal blood clotting profile
5. With wound or allergy over the treated acupoint
6. Unstable vital sign
7. Post major trauma

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) of dizziness | 20 minutes
  acupoints intervention of acupuncture or/and Far-Infrared heat-patch attachment